CLINICAL TRIAL: NCT04554147
Title: Patient-Provider-Community Health Worker Integrated Care Model: Use of an Innovative Mobile Health Intervention to Improve Hypertension Among African-Americans
Brief Title: Use of an Innovative Mobile Health Intervention to Improve Hypertension Among African-Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, LaPrincess C. Brewer, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-009247
Record Dates: First submitted 2020-07-12; First posted 2020-09-18 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: High Blood Pressure
Keywords: health disparities; mobile health; community health; African-Americans
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: This is a nonrandomized, single arm feasibility study testing the preliminary efficacy of an app-enhanced intervention with a patient-provider-community health worker triad to promote hypertension control among AA patients within FQHCs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAITH! App-enhanced Hypertension Intervention (Experimental): FAITH! HTN App: The program promotes HTN self-management through a 10-week education module series on HTN. Participants will follow each module weekly and use a wireless home BP monitor for self-tracking which syncs to the app. The app includes module quizzes, a BP tracking dashboard and a moderated sharing board to foster discussion on HTN management.
  Patient-Provider-CHW ICM. The patient-provider-CHW triad works together for personalized, collaborative goal setting. The patient will complete app modules, self-monitor BP, and engage with a sharing board integrating HTN topics. At weekly virtual visits (telephone or video), the CHW will record patient BPs, assist with addressing social determinants of health (SDOH) identified by the patient (eg, local community resources), and review HTN modules. The CHW will upload clinical/SDOH data to the patient electronic medical record (EMR) for FQHC care providers to review. This cycle will be completed weekly over the 10-week intervention.
  Interventions: Behavioral: FAITH! App-enhanced Hypertension Intervention

INTERVENTIONS:
Behavioral: FAITH! App-enhanced Hypertension Intervention — FAITH! HTN App: The program promotes HTN self-management through a 10-week education module series on HTN. Participants will follow each module weekly and use a wireless home BP monitor for self-tracking which syncs to the app. The app includes module quizzes, a BP tracking dashboard and a moderated sharing board to foster discussion on HTN management.
  Patient-Provider-CHW ICM. The patient-provider-CHW triad works together for personalized, collaborative goal setting. The patient will complete app modules, self-monitor BP, and engage with a sharing board integrating HTN topics. At weekly virtual visits (telephone or video), the CHW will record patient BPs, assist with addressing social determinants of health (SDOH) identified by the patient (eg, local community resources), and review HTN modules. The CHW will upload clinical/SDOH data to the patient electronic medical record (EMR) for FQHC care providers to review. This cycle will be completed weekly over the 10-week intervention.

SUMMARY:
The project objective is to test the feasibility of delivering health education and self-management support to African-American patients with uncontrolled hypertension (HTN) through a culturally-tailored smartphone application (app)-enhanced intervention within federally qualified health centers.

DETAILED DESCRIPTION:
The Fostering African-American Improvement in Total Health (FAITH!) Program at Mayo Clinic, a community-based cardiovascular (CV) health promotion initiative for African-Americans (AAs) will collaborate with the Minnesota Department of Health (MDH) Cardiovascular Health Unit and two federally qualified health centers (FQHCs) (NorthPoint Health & Wellness Center, Minneapolis, MN; Open Cities Health Center, St. Paul, MN) to integrate an innovative mobile health (mHealth) intervention (FAITH! HTN App) into clinical and community settings with the aim of improving blood pressure (BP) control.

The project objective is to test the feasibility of delivering health education and self-management support to African-American patients with uncontrolled hypertension (HTN) through a culturally-tailored smartphone application (app)-enhanced intervention within federally qualified health centers. This initiative is a component of a Centers for Disease Control and Prevention (CDC) effort to support state/local public health strategies to prevent and manage cardiovascular disease (CVD) in under-resourced populations disproportionately affected by CVD risk factors, such as HTN. Insights from the FAITH! Community Steering Committee (CSC) will also provide guidance to ensure project patient-centeredness. The investigators will incorporate strategies grounded in theoretical frameworks to ensure soundness of our intervention while tailoring it to meet the preferences and needs of an under-resourced population with multi-level barriers to HTN management.

Specific Aim 1:To assess app feasibility through participant intervention engagement (app education module completion, self-monitoring) and intervention satisfaction.

Specific Aim 2: To assess preliminary efficacy of the app by evaluating improvement in patient BP control (immediate, 3 months and 6 months post-intervention), CV health knowledge (via app self-assessments), and BP self-management (medication adherence).

Hypothesis:

The study hypothesis is that an app-based intervention will be feasible and demonstrate preliminary efficacy in improving uncontrolled HTN and health education among AA patients from baseline to post-intervention (immediate, 3 months and 6 months post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* African American race/ethnicity
* 18 years or older
* Receive primary care at one of the two partnering Federally Qualified Health Centers (FQHC) and intent to continue care there for next 6 months
* Uncontrolled HTN (defined as BP ≥140/90 mmHg [as per JNC7 Hypertension Guidelines68] at most recent outpatient evaluation, with or without BP medications)
* Documented diagnosis of HTN in EHR
* At least 1 office visit at one of the two partnering FQHCs in prior year
* Smartphone ownership (supporting iOS or Android Systems)

Exclusion Criteria:

* Unable to commit to participating in both focus groups (pre and post app refinement).
* Diagnosis of a serious medical condition or disability that would make participation difficult (i.e. visual or hearing impairment, mental disability that would preclude independent use of the app).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Blood pressure (systolic and diastolic, mmHg) | 0 months post intervention
  Change from baseline blood pressure.
Blood pressure (systolic and diastolic, mmHg) | 3 months post intervention
  Change from baseline blood pressure.
Blood pressure (systolic and diastolic, mmHg) | 6 months post intervention
  Change from baseline blood pressure.
Intervention Feasibility Measures - Participant Engagement with Self-Monitoring | Immediate post-intervention
  Participant engagement with weekly blood pressure tracking measured by number of times participant engaged with the blood pressure feature
Intervention Feasibility Measures - Participant Engagement with Self-Monitoring | Time Frame: 3 months post-intervention
  Participant engagement with weekly blood pressure tracking measured by number of times participant engaged with the blood pressure feature
Intervention Feasibility Measures - Participant Engagement with Self-Monitoring | Time Frame: 6 months post-intervention
  Participant engagement with weekly blood pressure tracking measured by number of times participant engaged with the blood pressure feature
HTN Self-Care Measures - Participant HTN self-care activities using the H-SCALE (Hypertension Self-Care Activity Level Effects) | Immediate post-intervention
  The 31-item instrument assess 6 HTN behavioral self-care activities recommended for optimal HTN management
HTN Self-Care Measures - Participant HTN self-care activities using the H-SCALE (Hypertension Self-Care Activity Level Effects) | 3 months post-intervention
  The 31-item instrument assess 6 HTN behavioral self-care activities recommended for optimal HTN management
HTN Self-Care Measures - Participant HTN self-care activities using the H-SCALE (Hypertension Self-Care Activity Level Effects) | 6 months post-intervention
  The 31-item instrument assess 6 HTN behavioral self-care activities recommended for optimal HTN management

SECONDARY OUTCOMES:
Preliminary Efficacy of Intervention - CV Health Knowledge as measured by module assessment scores | Immediate post intervention
  Change in percentage correct scores (pre- and post- self-assessments) for each education module by patient and as a conglomerate (mean) for all patients.
Social Determinants of Health (SDOH, PRAPARE (Protocol for Responding to and Addressing Patient Assets, Risks, and Experiences) tool) | Immediate post-intervention
  Change from baseline PRAPARE score. The PRAPARE assessment tool will be used to calculate a tally risk score indicating the cumulative number of SDOH risks a patient faces (including 15 SDOH domains).
Preliminary Efficacy of Intervention - BP Self-Management: Self-efficacy for HTN management | Immediate post-intervention
  Change from baseline score. Self-efficacy to change health behaviors to manage HTN as measured by a 5-item instrument.
Self Efficacy for Medication Adherence as measured by the MASES scale (medication adherence self-efficacy scale) | Immediate post-intervention
  Change from baseline score. The 13-item instrument assesses patients' confidence in their ability to take their BP medications in a variety of situations.

OTHER OUTCOMES:
Intervention Feasibility Measures - Participant Engagement with Sharing Board | Immediate post-intervention
  Participant engagement with sharing board measured by number of posts per week by each participant
Intervention Feasibility Measures - Participant Engagement with Sharing Board | 3 months post-intervention
  Participant engagement with sharing board measured by number of posts per month by each participant
Intervention Feasibility Measures - Participant Engagement with Sharing Board | 6 months post-intervention
  Participant engagement with sharing board measured by number of posts per month by each participant
Intervention Feasibility Measures - Participant Engagement with Modules | Immediate post-intervention
  Participant engagement with education modules measured by number of modules completed out of 10
Intervention Satisfaction Measures - Participant Satisfaction with FAITH! HTN App | Immediate post-intervention
  Participant satisfaction with FAITH! HTN App measured by the Health Information Technology Usability Evaluation Scale (Health-ITUES). 20 items are assessed, each on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree). A higher total sum indicates higher perceived usability of the technology.

CONTACTS AND LOCATIONS:
Overall Officials: LaPrincess C Brewer, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - North Point Health & Wellness Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Open Cities Health Center, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brewer LC, Jones C, Slusser JP, Pasha M, Lalika M, Chacon M, Takawira P, Shanedling S, Erickson P, Woods C, Krogman A, Ferdinand D, Underwood P, Cooper LA, Patten CA, Hayes SN. mHealth Intervention for Promoting Hypertension Self-management Among African American Patients Receiving Care at a Community Health Center: Formative Evaluation of the FAITH! Hypertension App. JMIR Form Res. 2023 Jun 16;7:e45061. doi: 10.2196/45061. PMID 37115658
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT04554147/ICF_000.pdf